CLINICAL TRIAL: NCT05561712
Title: Method Optimization for the Quantification of the NAD (Nicotinamide Adenine Dinucleotide) Metabolome in Human Whole Blood, Plasma, and Urine, and Evaluation of Baseline Inter and Intra-subject Variability
Brief Title: Method Optimization for the Quantification of the NAD
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 2112NR
Record Dates: First submitted 2022-03-03; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: NAD
Keywords: NAD quantification in blood and urine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Laboratory method validation — Test several sampling conditions

SUMMARY:
Method optimization for the quantification of the NAD metabolome in human whole blood, and evaluation of baseline inter and intra-subject variability.

DETAILED DESCRIPTION:
Whole blood from healthy participants will be collected to optimize analytical method based on liquid chromatography tandem mass spectrometry (LC-MS/MS) for the analysis of the NAD metabolome in biological samples. Parameters such as collection volume and anti-coagulants will be investigated for optimal quantification. Moreover, inter- and intra-subject variability of NAD metabolite levels in whole blood will be evaluated. Plasma and urine will also collected for method development and variability measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women (based on anamnesis),
2. Age between 18 and 55 years,
3. Body Mass Index (BMI) = weight (kg) / height (m)2 between 18.5 to 28 kg/m2.

Exclusion Criteria:

1. Pregnant or lactating women
2. Sick or with a strong cold
3. With vitamin B3 supplementations or under low carbohydrate of ketogenic diet
4. Under prescribed chronic medication, except contraceptive pill.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Comparison of NAD metabolite concentrations in whole blood, collected with different tubes and anticoagulants. | through study completion, an average of 1 year
  NAD metabolites in whole blood will be quantified by liquid chromatography-tandem

SECONDARY OUTCOMES:
Estimation of inter- and intra-subject variabilities of NAD metabolites in whole blood | through study completion, an average of 1 year
  Descriptive estimates of the inter and intra subjects variances will be calculated with the standard formulas.
Validation of the method for a set of NAD metabolites in plasma and urine (including determination of Limit Of Detection-LOD, Limit Of Quantification- LOQ). | through study completion, an average of 1 year
  NAD metabolites in urine and in blood will be quantified to enable to measure several validation parameters, such as intra and interday precision, LOD, LOQ, r2.

CONTACTS AND LOCATIONS:
Overall Officials: Cuenoud Bernard, Study Director — Nestle Health Science
Locations (1):
- Clinical Innovation Lab., Lausanne, Switzerland